CLINICAL TRIAL: NCT01098851
Title: Saturation Pattern Detection Prevalence Study Protocol
Brief Title: Oxygen Saturation Monitoring During Surgery
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COV-MO-PO-1000
Record Dates: First submitted 2010-03-31; First posted 2010-04-05 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Pulse Oximetry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea: Surgery patients at high risk for Obstructive Sleep Apnea
- Surgery Patients: Surgery patients at low risk for Obstructive Sleep Apnea

SUMMARY:
Patients with Obstructive Sleep Apnea (OSA) have cyclical patterns of lower blood oxygen during sleep because of repeated episodes of upper airway obstruction that cause their breathing to stop. When these patients have surgery, anesthetic drugs may worsen these patterns of lower blood oxygen. This study monitors ten patients at high risk for OSA and ten patients at low risk for OSA during surgery. Patterns of lower oxygen saturations should arise in the high risk group but not the low risk group.

DETAILED DESCRIPTION:
Patients with Obstructive Sleep Apnea (OSA) have episodes of upper airway obstruction during sleep which have been shown to be accompanied by multiple oxygen desaturations followed by short recovery intervals until rising PaCO2 causes sleep disruption/rescue arousal. In the postoperative and conscious sedation arena, these patterns can deteriorate from a stable pattern to a severely unstable pattern which may go unrecognized and lead to an adverse event (respiratory/cardiac arrest; death).

Anesthesia and the higher consumption of analgesics produce a profound reduction in pharyngeal tone, a dampening of both chemoreceptor sensitivity and arousal/rescue response. Thus the first 48 hours post operatively presents a vulnerable period. Respiratory disturbances are more prominent - respiratory arrest and hypopnea being the main adverse occurrences during this period.

An algorithm has been developed that monitors saturation and indicates repetitive reductions in airflow through the upper airway and into the lungs. Presence of this pattern in the procedural sedation patient population has not been tested for its prevalence. This study will monitor patients during surgery to determine if this pattern occurs in this hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 21 years
* Patients scheduled for a procedure that requires analgesia and/or sedation by any route (intravenous, intramuscular, oral, epidural or intrathecal).
* Patients with an anticipated length of sedation greater than or equal to one hour.
* Patients in the ASA category I through III.
* Patients who only receive propofol, benzodiazepines, and opioids.

Exclusion Criteria:

* Age less than 21 years
* Patients whose room air oxygen saturation is <90%
* Patients receiving post-operative positive airway pressure support
* Previous allergic/contact reactions to adhesives
* CHF
* Moderate or severe valvular disease
* TIA/CVA
* Carotid stenosis or endarterectomy
* Anemia (HCT if available < 30%)
* Pulmonary hypertension
* Dialysis
* Pregnancy
* Patients unable to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Mecca, MD, Study Chair — Medtronic - MITG
Locations (1):
- Avista Adventist Hospital, Louisville, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from July through November 2009 in the medical clinic who were scheduled for surgery that required procedural sedation.
Period: Overall Study
Arm/Group | Obstructive Sleep Apnea | Surgery Patients
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Equipment failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obstructive Sleep Apnea | Surgery Patients | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10) | 36 (7) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Saturation Pattern Detection (SPD) Indicative of Repetitive Reductions in Air Flow
Description: Saturation Pattern Detection (SPD) is the pattern of oxygen saturation values plotted against time that occurs when patients have cyclical reduced air movement during breathing. Their blood oxygen level decreases and increases as they slow and increase their breathing.
Time Frame: 3 hours
Measure: Number; unit: Participants
Arm/Group | Obstructive Sleep Apnea | Surgery Patients
Number analyzed (Participants) | 11 | 10
Participants | 4 | 0

2. Primary Outcome: Number of Participants Requiring Airway Support
Description: Drugs during surgery may cause the throat to relax and block breathing. To treat this, the caregiver administers airway support. Airway support is moving the jaw forward, inserting a plastic tube (nasal-oral airway) or applying a mask with positive pressure.
Time Frame: 3 hours
Measure: Number; unit: Participants
Arm/Group | Obstructive Sleep Apnea | Surgery Patients
Number analyzed (Participants) | 11 | 10
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Obstructive Sleep Apnea | Surgery Patients
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less